CLINICAL TRIAL: NCT01176448
Title: A Comparison Evaluation of Fractional Laser Therapy and Dermabrasion for Scar Revision
Brief Title: Laser Resurfacing Versus Dermabrasion for Scar Revision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1001M75732-2
Record Dates: First submitted 2010-06-21; First posted 2010-08-06 (Estimated); Results first posted 2013-06-27 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Cicatrix; Dermabrasion; Coagulation, Laser
Keywords: Cicatrix; Dermabrasion; Coagulation, Laser
MeSH Terms: conditions — Cicatrix; Thrombosis | interventions — Dermabrasion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fractionated laser (Experimental): This Arm is the section of scar that will be treated with Fractionated Laser
  Interventions: Device: Fractionated laser
- Dermabrasion (Active Comparator): Dermabrasion is the gold standard for scar resurfacing and will be used as the control against which Fractionated Laser is compared.
  Interventions: Device: Dermabrasion

INTERVENTIONS:
Device: Fractionated laser — Fractionated laser in the form of the Re:Pair CO2 laser manufactured by Solta Medical.
  Arms: Fractionated laser
Device: Dermabrasion — Diamond Fraise Dermabrasion will be performed in standard fashion down to papillary dermis.
  Arms: Dermabrasion

SUMMARY:
Dermabrasion has been the historical standard used for resurfacing scars on the skin. Recently, fractionated laser therapy has been FDA approved for scar resurfacing. This study intends to compare dermabrasion versus fractionated laser therapy for scar resurfacing.

ELIGIBILITY:
Inclusion Criteria:

* Post-surgical or post traumatic scar on face or scalp.
* Age 18 or older
* Able to read and comprehend English
* Willing to follow treatment schedule and post treatment care requirements
* Signed the informed consent form
* Fitzpatrick skin type I-III

Exclusion Criteria:

* known photosensitivity
* Taken any medications known to induce photosensitivity in previous three months
* Taken Accutane within past 12 months
* Pregnant or nursing
* Currently on topical or oral antibiotics
* Immunocompromised status
* Skin type IV or greater

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Christophel, MD, Principal Investigator — University of Minnesota
Locations (1):
- Zel Skin and Laser, Edina, Minnesota, United States

REFERENCES:
- [Derived] Jared Christophel J, Elm C, Endrizzi BT, Hilger PA, Zelickson B. A randomized controlled trial of fractional laser therapy and dermabrasion for scar resurfacing. Dermatol Surg. 2012 Apr;38(4):595-602. doi: 10.1111/j.1524-4725.2011.02283.x. Epub 2012 Jan 23. PMID 22268699

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients aged 18 and older were recruited from a reconstructive surgical practice. Preference was given to patients who had undergone interpolated axial flaps (e.g., forehead flaps) because this allowed treatment of two different scars on a single patient.
Groups:
- Patients With Scars: 12 long scars were recruited for individual study. Only 6 patients were needed as each patient had two separate scars to be studied. Each scar was divided in half, and the halves randomized to fractionated laser resurfacing or dermabrasion.
  The half of the scar randomized to fractionated CO2 laser was treated first. The Re:Pair CO2 laser was used, with a fluence of 40 mJ and a treatment level of 8 (Solta Medical Inc., Hayward, CA). Four passes of the laser were used in total, with two in the orthogonal direction. A standard diamond fraise dermabrader was used on the area painted with gentian violet down through the dermal-epidermal junction. Dermabrasion was performed until a uniform area of punctate bleeding was obtained, and the edges were feathered into the surrounding epidermis.
Period: Overall Study
Arm/Group | Patients With Scars
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 12 long scars were recruited for individual study. Only 6 patients were needed as each patient had two separate scars to be studied. Each scar was divided in half, and the halves randomized to fractionated laser resurfacing or dermabrasion.
Groups:
- Patients With Scars: 12 individual scars on 6 patients were treated. Each scar was divided in half, and the halves randomized to either fractionated laser resurfacing or dermabrasion.
Arm/Group | Patients With Scars
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Safey Data Score Based on Ordinal Ratings of Erythema, Edema, Bleeding, Eschar After Resurfacing
Description: Erythema, edema, bleeding, and eschar after resurfacing were used as indicators of safety. Each was judged based on a 4 point ordinal scale 0=absent, 1=mild, 2=moderate, 3=severe.
Time Frame: Day 0, Week1, Month 1
Population: Each scar was divided in half and the halves randomized to either Fractionated Laser treatment or Dermabrasion.
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: Scars
Arm/Group | Fractionated Laser | Dermabrasion
Number analyzed (Participants) | 6 | 6
Number analyzed (Scars) | 12 | 12
units on a scale
  Erythema Day 0 | 1.33 (0.49) | 3.00 (0)
  Edema Day 0 | 0 (0) | 0 (0)
  Bleeding Day 0 | 1.08 (0.29) | 2.0 (0)
  Eschar Day 0 | 0 (0) | 0 (0)
  Erythema Week 1 | 0.75 (0.45) | 1.50 (0.52)
  Edema Week 1 | 0.17 (0.39) | 0.50 (0.52)
  Bleeding Week 1 | 0 (0) | 0 (0)
  Eschar Week 1 | 0.08 (0.29) | 0.92 (0.79)
  Erythema Month 1 | 0.38 (0.52) | 1.25 (1.04)
  Edema Month 1 | 0 (0) | 0 (0)
  Bleeding Month 1 | 0 (0) | 0 (0)
  Eschar Month 1 | 0 (0) | 0 (0)

2. Secondary Outcome: Visual Analog Scale for Assessing Scar Improvement.
Description: Visual Analog Scale for assessing scar improvement. 0 : Worsening or no improvement
  1. : 1-25% improvement
  2. : 26-50% improvement
  3. : 51-75% improvement
  4. : 76-100% improvement
Time Frame: 3 months
Population: With 12 pairs of scars gave a 95% probability to detect a treatment difference at a two sided 0.05 significance level if a significant difference between treatments is 1.5 units (based on a 0
  -4 scale as mentioned above). This is based on the assumption that the within-patient standard deviation of the response variable is 0.5 units.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Scar Halves
Groups:
- Fractionated Laser: This Arm is the section of scar that will be treated with Fractionated Laser. 6 patients had 12 scars treated (2 scars per patient.
- Dermabrasion: Dermabrasion is the gold standard for scar resurfacing and will be used as the control against which Fractionated Laser is compared. 6 patients had 12 scars treated (2 scars per patient.
Arm/Group | Fractionated Laser | Dermabrasion
Number analyzed (Participants) | 6 | 6
Number analyzed (Scar Halves) | 12 | 12
units on a scale | 1.53 (.59) | 1.49 (.39)
Statistical Analysis 1: Comparison: Fractionated Laser vs Dermabrasion; efficacy outcomes analyzed by 3 surgeons blinded to the treatment and scars evaluated by halves comparing pre-treatment photos to 3-month photos and given a score on the quartile scale described in table 1. The ordinal rater scores of each evaluator were then averaged, and Wilcoxon Signed Ranks performed on the group's scores. (table 5) There were 4 Fraxel winners, 4 Dermabrasion winners, and 4 ties. There was a p value of 0.77 indicating no significant difference between the categories; Test type: Non-Inferiority or Equivalence — With 12 scars (or pairs to compare), our power calculation had a 95 percent probability that the study will detect a treatment difference at a two-sided 0.05 percent significance level, if a significant difference between treatments is 1.5 units (based on a 0-4 scale as mentioned above). This is based on the assumption that the within-patient standard deviation of the response variable is 0.5 units; p = .77, Wilcoxon (Mann-Whitney) — Appropriately powered, this study failed to reject the null hypothesis that fraxel achieves a similar cosmetic result at 3 months when compared to dermabrasion

ADVERSE EVENTS:
Arm/Group | Fractionated Laser | Dermabrasion
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No